CLINICAL TRIAL: NCT03972371
Title: The ProVerum First in Man PROVE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProVerum Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-001
Record Dates: First submitted 2019-05-17; First posted 2019-06-03 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomised, single centre, safety and feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): The ProVee Urethral Expander is implanted into the prostatic urethra to treat BPH symptoms
  Interventions: Device: The ProVee Urethral Expander System

INTERVENTIONS:
Device: The ProVee Urethral Expander System — The ProVee Urethral Expander System is supplied as a single use, sterile device and consists of a nitinol expander implant and custom implant delivery system. The delivery system is designed to allow the implant to be deployed under direct vision.
  Other Names: The ProVee Expander

SUMMARY:
A clinical evaluation to assess the safety and performance of the ProVeeTM Urethral Expander System, designed to alleviate the symptoms of Benign Prostatic Hyperplasia (BPH).

ELIGIBILITY:
Inclusion Criteria:

* Males ≥ 50 years of age
* Moderate-to-severe symptomatic BPH
* IPSS of > 15
* Peak urinary flow rate (Qmax) of <12 mL/s
* Prostate volume of ≥ 30 and ≤80 cc
* Prostatic urethral lengths ≥ 4cm

Exclusion Criteria:

* A prostatic urethral length of less than 4cm
* A prostatic volume <30cc or >80cc
* An obstructing intravesical prostatic median lobe
* Urinary incontinence due to an incompetent external sphincter
* Urethral pathologies that may prevent insertion of delivery system
* A current symptomatic urinary tract infection
* Current significant visible haematuria
* Patients with known allergy to nickel or titanium
* History of significant medical co-morbidity or prior surgery that may confound the results of the Study
* Another medical condition that would pose an unacceptable patient risk
* Known or suspected urological condition that may affected voiding function
* Neurogenic bladder and/or sphincter abnormalities
* Patients with cognitive disabilities unable to understand and give informed consent to the research study

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 10 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Deployment of the Implant | Immediately after the implant deployment procedure
  Successful deployment of the implant from the delivery system in the target location within the prostatic urethra, as assessed with post deployment endoscopy
Expansion of the Implant | Within 24 hours of the implant deployment procedure
  Successful deployment of the implant from the delivery system in the target location within the prostatic urethra, as assessed with post deployment CT

SECONDARY OUTCOMES:
Rate of complications e.g. difficulty with urination, related to the implant use peri-procedurally and in the immediate follow up period | Immediately after the implant deployment procedure, within 24 hours
Rate of complications e.g. pain, difficulty with urination, related to the implant throughout the follow-up period of 2 years | 2 years
Preliminary assessment of the effectiveness of the procedure in alleviating LUTS voiding symptoms | 2 years
  Change in symptom score using the Improvement in International Prostate Symptom Score and Quality of Life score instrument within the 2 year follow up period
Preliminary assessment of the effectiveness of the procedure in improving urinary flow | 2 years
  Change in Qmax measurement within the 2 year follow up period

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Melbourne Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No